CLINICAL TRIAL: NCT02765035
Title: A Randomized, Blinded, Cross-over Trial to Evaluate the Safety, Functional Mobility and Satisfaction of the Microprocessor Controlled Prosthetic Knee Component C-Leg 4 in Transfemoral Amputees
Brief Title: C-Leg 3 and C-Leg 4 Study in Transfemoral Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PD-PS00120010A-001
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C-Leg 3, then C-Leg 4 (Experimental): Participants are first fitted with a C-Leg 3, receive physical therapy, acclimate for 90 days and are then assessed in the clinic. They then receive a C-Leg 4, receive additional physical therapy and acclimate for 30 days after which they are again assessed in the clinic.
  Interventions: Device: C-Leg 4; Device: C-Leg 3
- C-Leg 4, then C-Leg 3 (Experimental): Participants are first fitted with a C-Leg 4, receive physical therapy, acclimate for 90 days and are then assessed in the clinic. They then receive a C-Leg 3, receive additional physical therapy and acclimate for 30 days after which they are again assessed in the clinic.
  Interventions: Device: C-Leg 4; Device: C-Leg 3

INTERVENTIONS:
Device: C-Leg 4 — Microprocessor Controlled Knee
Device: C-Leg 3 — Microprocessor Controlled Knee

SUMMARY:
The aim of this post-market study is to confirm that the microprocessor controlled prosthetic knee components (C-Leg 3 and C-Leg 4) in comparison to mechanical knee joints can bring additional benefit to the users primarily on level walking and secondarily in safety, stair and hill mobility, activities of daily living, satisfaction and preference.

DETAILED DESCRIPTION:
During the last two decades many microprocessor controlled knee joints (MPK) appeared on the market.The newly developed C-Leg 4 aims to provide improved standing function while in the same time offering technology of knee´s previous version (C-Leg 3). Since added functional benefit of a knee joint cannot be anticipated just due to the fact that the knee is controlled by the microprocessor, the aim of this post-market study is to evaluate the safety, functional mobility and satisfaction of the microprocessor controlled prosthetic knee components C-Leg 3 and C-Leg 4 in comparison to mechanical knee joints. Additional goal is to improve the methodological quality of research conducted in the field.

ELIGIBILITY:
Inclusion Criteria:

* Person is >18 years old.
* Person is a unilateral transfemoral or knee-disarticulation amputee with stabilized residual limb.
* Person is a K2, K3 or K4 ambulator based on Medicare Functional Classification Level (MFCL).
* Person is currently fitted with a prosthesis using a non-microprocessor controlled prosthetic knee for at least 6 months.
* Person was never fitted with microprocessor controlled prosthetic knee joint.
* Person is willing and able to independently provide informed consent.
* Person is willing to comply with study procedures.
* Person wears prosthesis daily and ≥ 8 hours/day.
* Person is walking on average 1km/day.
* Person is walking not slower than 3km/h (~0.8m/s) (based on 10m walk test conducted during recruiting).
* Person is walking on level ground in a step over step manner.

Exclusion Criteria:

* Person is under 18 years of age.
* Person who weighs more than 136kg.
* Person who weighs less than 50kg.
* Person who is pregnant.
* Person has a history of chronic skin breakdown on the residual limb.
* Person has conditions that would prevent participation and pose increased risk (e.g. unstable cardiovascular conditions that preclude physical activity such as walking).
* Person falls ≥ once a week due to the reasons that could not be corrected by the new prosthesis (for ex. problems with vestibular system).
* Person is using under arm axillary crutches or walker.
* Person in an emergency, life threatening situation.
* Person is unwilling/unable to follow instructions.
* Person who is not available to follow the entire study protocol.
* Person who is participating in another study or intends to participate in another study during this study duration.
* Person who cannot personally provide their consent.
* Person who is not wearing prosthesis 8hours/day on average.
* Person who has a score on 10m walk test less than 3km/h (~0.8m/s) (based on 10m walk test conducted during recruiting).
* Person who walks on average less than 1km per day.
* Person who is not able to walk on level ground in a step over step manner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-04; Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Domayer, Prim.Dr., Principal Investigator — Orthopedic Rehabilitation Center
Locations (2):
- Orthopedic Rehabilitation Center SKA Zicksee, Sankt Andrä am Zicksee, Burgenland, Austria
- University Leuven, Pellenberg, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data for primary and secondary outcome measures will be made available within one year of study completion.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 subjects were excluded from the study prior to randomization: 3 subjects had adverse events, 1 subject could not be fitted with the intervention device due to anthropomorphic characteristics, and 1 subject withdrew due to a change in work situation.
Groups:
- C-Leg 3, Then C-Leg 4: The participants were first fitted with C-Leg 3 and allowed to accommodate for up to 90 days after which they were assessed. Then they crossed over to be fitted with the C-Leg 4 and allowed to accommodate for 30 days after which they were assessed.
- C-Leg 4, Then C-Leg 3: The participants were first fitted with C-Leg 4 and allowed to accommodate for up to 90 days after which they were assessed. Then they crossed over to be fitted with the C-Leg 3 and allowed to accommodate for 30 days after which they were assessed.
Period: First Intervention (90 Days)
Arm/Group | C-Leg 3, Then C-Leg 4 | C-Leg 4, Then C-Leg 3
Started | 5 | 8
Completed | 4 | 7
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Second Intervention (30 Days)
Arm/Group | C-Leg 3, Then C-Leg 4 | C-Leg 4, Then C-Leg 3
Started | 4 | 7
Completed | 2 | 5
Not Completed | 2 | 2
Not completed — Protocol Violation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C-Leg 3, Then C-Leg 4 | C-Leg 4, Then C-Leg 3 | Total
Number analyzed (Participants) | 5 | 8 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (4.95) | 58.5 (12.2) | 60.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 5 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 2 | 2 | 5
  Belgium | 3 | 6 | 8
Height [Mean (Standard Deviation); unit: cm] | 177.4 (7.54) | 172.13 (9.40) | 174.15 (8.81)
Weight [Mean (Standard Deviation); unit: kg] | 74.4 (12.4) | 73.9 (14.4) | 74.1 (13.1)
Time since amputation [Mean (Standard Deviation); unit: years] | 21.8 (23.6) | 23.0 (14.9) | 22.54 (17.74)
Amputation side [Count of Participants; unit: Participants]
  left | 1 | 3 | 4
  right | 4 | 5 | 9
Amputation type [Count of Participants; unit: Participants]
  Transfemoral | 0 | 4 | 4
  Knee disarticulation | 5 | 4 | 9
Medicare Functional Classification Level (MFCL) [Count of Participants; unit: Participants] — The Medicare Functional Classification Level (MFCL) was adopted in 1995 by the US Centers for Medicare and Medicaid Services using 5 levels for classifying functional mobility and rehabilitation potential of individuals with lower limb loss. Level 0 does not have the ability or potential to ambulate or transfer safely. Level 1 is a household ambulator. Level 2 is a limited community ambulator. Level 3 is a community ambulator, and Level 4 has higher prosthetic demands typical of the child, active adult or athlete.
  Participants
    2 | 1 | 1 | 2
    3 | 4 | 6 | 10
    4 | 0 | 1 | 1
Current knee prosthesis (NMPK) [Count of Participants; unit: Participants]
  3R106 | 1 | 3 | 4
  3R15 | 0 | 1 | 1
  3R60 | 2 | 1 | 3
  3R80 | 2 | 1 | 3
  Polycentric | 0 | 1 | 1
  Multiaxial | 0 | 1 | 1
Amputation cause [Count of Participants; unit: Participants]
  cancer | 1 | 5 | 6
  infection | 1 | 1 | 2
  trauma | 1 | 1 | 2
  vascular disease | 2 | 1 | 3
Hours of wearing prosthesis per day [Mean (Standard Deviation); unit: hours] | 12.4 (2.6) | 12.4 (2.7) | 12.4 (2.6)
Distance covered per day [Mean (Standard Deviation); unit: km] | 3.6 (2.1) | 3.25 (1.5) | 3.38 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in 6 Minute Gait Test
Description: A measure of walking endurance, the distance walked in meters after 6 minutes.
Time Frame: Baseline and after acclimation period (30-90 days after fitting)
Measure: Mean (Standard Deviation); unit: meters
Groups:
- C-Leg 3: The participants wearing a C-Leg 3 either in the first fitting (after max 90 days of acclimation) or the second fitting (after 30 days acclimation)
- C-Leg 4: The participants wearing a C-Leg 4 either in the first fitting (after max 90 days of acclimation) or the second fitting (after 30 days acclimation)
Arm/Group | C-Leg 3 | C-Leg 4
Number analyzed (Participants) | 7 | 7
meters
  Baseline | 380.4 (69.66) | 380.4 (69.66)
  Change from Baseline after accommodation | 35.9 (20.26) | 26.7 (33.87)
Statistical Analysis 1: Comparison: C-Leg 3; C-Leg 3 vs. NMPK (Baseline); Test type: Superiority; p = 0.01, t-test, 1 sided
Statistical Analysis 2: Comparison: C-Leg 4; C-Leg 4 vs. NMPK (Baseline); Test type: Superiority; p = 0.04, t-test, 1 sided

2. Secondary Outcome: Change in 10 Meter Gait Test
Description: Average gait speed over middle 6 meters of a 10-meter course at both self-selected and fastest safe walking speeds
Time Frame: Baseline and after acclimation period (30-90 days after fitting)
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | C-Leg 3 | C-Leg 4
Number analyzed (Participants) | 7 | 7
meters per second
  SSWS at Baseline | 1.11 (0.168) | 1.11 (0.168)
  SSWS after acclimation | 0.00 (0.06) | -0.25 (0.14)
  FWS at Baseline | 1.36 (0.262) | 1.36 (0.262)
  FWS after acclimation | 0.21 (0.15) | -0.03 (0.08)

3. Secondary Outcome: Change in Stairs Assessment Index (SAI)
Description: Participants are scored on a 14-level scale for independence, technique and step length for ascending and descending a 12-step ADA-compliant stairwell. The maximum score is 13 and the minimum 0. Higher scores indicate greater independence. Time to descend stairs was also recorded.
Time Frame: Baseline and after acclimation period (30-90 days after fitting)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | C-Leg 3 | C-Leg 4
Number analyzed (Participants) | 7 | 7
score on a scale
  Baseline SAI (Ascent) | 5 (2.6) | 5 (2.6)
  Change in SAI (Ascent) after fitting and acclimation | -0.6 (1.5) | 0.0 (0.0)
  Baseline SAI (Descent) | 4 (1.6) | 4 (1.6)
  Change in SAI (Descent) after fitting and acclimation | 5.9 (3.2) | 5.7 (2.9)
  Baseline time to descent stairs | 12.7 (3.95) | 12.7 (3.95)
  Change in time to descent stairs after fitting and acclimation | -2.1 (1.7) | -3.1 (2.0)

4. Secondary Outcome: Change in Hill Assessment Index (HAI)
Description: Participants are scored on a 12-level scale for independence, technique and step length for descending a 5m, 5-degree downgrade hill at self selected speed. The maximum score is 11 and the minimum 0. Higher scores indicate greater independence. Time to descend the hill was also recorded.
Time Frame: Baseline and after acclimation period (30-90 days after fitting)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | C-Leg 3 | C-Leg 4
Number analyzed (Participants) | 7 | 7
score on a scale
  Baseline HAI (Ascent) | 8.4 (2.5) | 8.4 (2.5)
  Change in HAI (Ascent) after fitting and acclimation | 1.9 (2.0) | 1.1 (1.3)
  Baseline HAI (Descent) | 7.9 (2.8) | 7.9 (2.8)
  Change in HAI (Descent) after fitting and acclimation | 1.9 (2.0) | 0.9 (2.7)
  Baseline Descent Time | 6.6 (2.5) | 6.6 (2.5)
  Change in Descent Time after fitting and acclimation | -0.9 (1.3) | -0.4 (1.4)

5. Secondary Outcome: Change in Four Step Square Test (FSST)
Description: Time to complete a stepping sequence through 4 squares as quickly as possible. The test involves stepping forward, backward and sideways to the left and right while face the same direction.
Time Frame: Baseline and after acclimation period (30-90 days after fitting)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | C-Leg 3 | C-Leg 4
Number analyzed (Participants) | 7 | 7
seconds
  Baseline FSST | 13.5 (3.92) | 13.5 (3.92)
  FSST after fitting and acclimation | -2.6 (1.18) | -2.4 (1.77)

6. Secondary Outcome: Change in Activities-specific Balance Confidence (ABC) Scale
Description: Assessment of patient-perceived balance confidence for 16 activities of daily living. For each activity, subjects rate their level of confidence in doing the activity without losing their balance or becoming unsteady on a scale from 0% to 100%, with 100% being the highest level of confidence. The total score for the ABC scale is an average of all activity scores.
Time Frame: Baseline and after acclimation period (30-90 days after fitting)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | C-Leg 3 | C-Leg 4
Number analyzed (Participants) | 7 | 7
score on a scale
  Baseline ABC | 72.4 (9.73) | 72.4 (9.73)
  Change in ABC after fitting and acclimation | 1.4 (7.83) | 2.7 (8.75)

7. Secondary Outcome: Change in Prosthetic Limb Users Survey of Mobility (PLUS-M)
Description: The PLUS-M 12-item short form is a valid and reliable self-reported measure for the mobility of adults with lower limb amputations. PLUS-M asks about the patient's ability to perform simple and complex tasks. Higher PLUS-M scores correspond with greater mobility. T-scores range from 21.8 to 71.4. A T-score has a mean of 50 and a standard deviation (SD) of 10. A PLUS-M T-score of 50 represents the mean mobility reported by the development sample (i.e., people with unilateral amputation).
Time Frame: Baseline and after acclimation period (30-90 days after fitting)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | C-Leg 3 | C-Leg 4
Number analyzed (Participants) | 7 | 7
T-score
  Baseline PLUS-M T-Score | 50.0 (6.64) | 50 (6.64)
  Change in PLUS T-Score after fitting and acclimation | 0.6 (3.3) | 0.8 (3.27)

8. Secondary Outcome: Change in Amputee Body Image Scale (ABIS)
Description: The ABIS assesses how an amputee perceives and feels about his or her body experience. The scale addresses several different domains, including: 1) body appearance; 2) body function; 3effective distress; and 4) behavioral avoidance in social situations. The scale produces scores that range from 1 to 100, with low scores indicating the relative absence of a body image concern and higher scores indicating the presence of a more serious body-image concern.
Time Frame: Baseline and after acclimation period (30-90 days after fitting)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | C-Leg 3 | C-Leg 4
Number analyzed (Participants) | 7 | 7
score on a scale
  Baseline ABIS | 55.1 (13.01) | 55.1 (13.01)
  Change in ABIS after fitting and acclimation | 1.9 (7.34) | -0.4 (6.97)

9. Secondary Outcome: Change in Number of Stumbles and Falls
Description: Stumbles and falls in the previous 30 days for each studied device based on records in a subject log book. At baseline, users were asked to recall the number of stumbles and falls in the previous 30 days.
Time Frame: Baseline and after acclimation period (30-90 days after fitting)
Measure: Mean (Standard Deviation); unit: number of stumbles or falls
Arm/Group | C-Leg 3 | C-Leg 4
Number analyzed (Participants) | 7 | 7
number of stumbles or falls
  Baseline number of stumbles | 3.3 (4.07) | 3.3 (4.07)
  Change in number of stumbles after fitting and acclimation | -0.3 (2.56) | -0.3 (2.29)
  Baseline number of falls | 1.0 (1.53) | 1.0 (1.53)
  Change in number of falls after fitting and acclimation | -0.6 (1.62) | -0.1 (1.77)

10. Secondary Outcome: Preference of the Knee (Percentage of Subjects That Preferred Each Studied Knee)
Description: The user´s knee preference is assessed with the question: "Which prosthesis do you prefer?"
Time Frame: At 3rd study visit after having been fitted and acclimatized to each of the study devices
Population: All subjects with preference data that completed the study were included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: All subjects were ask which knee they preferred after having been fitted and acclimatized to each (C-Leg 3, C-Leg 4 and the NMPK)
Arm/Group | All Subjects
Number analyzed (Participants) | 11
Participants
  Number preferring the C-Leg 4 | 7
  Number preferring the C-Leg 3 | 3
  Number preferring the NMPK | 1

ADVERSE EVENTS:
Time Frame: 36-40 weeks
Arm/Group | C-Leg 3 | C-Leg 4
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 3/13 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C-Leg 3 (N=13) | C-Leg 4 (N=13)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Residual limb pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
From 11 subjects that participated in the study, only 7 followed protocol. From post-hoc power analysis, 22 subjects would be required for 80% power to detect a difference of 35.9m (standard deviation = 30.3m) in the 6MWT.

Patients were aware that a walking speed of greater than 0.8 m/s was a prerequisite for study participation, which could have lead to bias (elevated baseline measurement) and explain the small change in observed walking speed with C-Leg 3 and C-Leg 4 compared to baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT02765035/Prot_SAP_000.pdf